CLINICAL TRIAL: NCT01522222
Title: Effect of Continuous Mechanical Ventilation During Cardiopulmonary Bypass on The Lung Mechanics: A Prospective Evaluation
Brief Title: Study to Determine if Using Ventilation During Open Heart Surgery Improves Lung Outcomes
Acronym: PEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aurora BayCare Medical Center (Other)
Responsible Party: Principal Investigator, Raul Mendoza-Ayala, Pulmonologist, Aurora BayCare Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PEEP
Record Dates: First submitted 2012-01-24; First posted 2012-01-31 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Coronary Artery Disease; Heart Failure
Keywords: cardiopulmonary bypass surgery; CABG; PEEP
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): half of the study subjects will receive standard of care during their open heart surgery.
- Treatment (Experimental): half of the study subjects will receive the prescribed ventilatory support during open heart surgery.
  Interventions: Procedure: continuous, mechanical ventilatory support

INTERVENTIONS:
Procedure: continuous, mechanical ventilatory support — Those in the treatment group will receive ventilation, intermittent positive pressure ventilation, while their heart is arrested. The subjects will have their lungs ventilated six times per minute with a tidal volume equal to 7-10 milliliters per kilogram. This range, when combined with a consistent PEEP of 5cm of water pressure, will allow for the peak inspiratory pressure to be maintained at or below 40cm of water pressure. In addition, the FIO2 will remain consistent at the same level that was needed to maintain the pulse oximetry at 94% as well as the end-tidal CO2 at 35mmHg.
  Arms: Treatment

SUMMARY:
To demonstrate that using continuous mechanical lung ventilatory support in combination with Positive End Expiratory Pressure (PEEP)during open heart surgery will improve lung function and decrease lung complications after surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, blinded study with a control group. The study group will receive mechanical ventilatory support during CBB, which consists of a preset/predetermined tidal volume, respiratory rate, positive pressure at the end of expiration and FIO2. The control group will receive CPB without additional mechanical ventilatory support during surgery, which at present is the standard of care.

The difference between the study and the control group will occur during the time the heart is arrested and the lungs, under present standard of care, are no longer ventilated. It is at this point in time that those in the study group will continue to receive ventilation, intermittent positive pressure ventilation, while their heart is arrested. The subjects will have their lungs ventilated six times per minute with a tidal volume equal to 7-10 milliliters per kilogram. This range, when combined with a consistent PEEP of 5cm of water pressure, will allow for the peak inspiratory pressure to be maintained at or below 40cm of water pressure. In addition, the FIO2 will remain consistent at the same level that was needed to maintain the pulse oximetry at 94% as well as the end-tidal CO2 at 35mmHg. The values mentioned for this study have been chosen based on not only investigator preference, but also on what is considered "minimally necessary" to prevent atelectasis. Multiple studies have been done utilizing PEEP at 5 and 10 cm of water pressure. With the exception of the potential for mechanical ventilation during the CBP, the care of the subject, regardless of the group randomized into, will be the same. We will in all other aspects continue to utilize the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* any patient of any gender, any age with known coronary artery disease that will undergo elective Coronary Artery Bypass Grafting (CABG) and will require CPB as part of his/her operative technique.

Exclusion Criteria:

* documented ejection fraction (either by echocardiogram or by cardiac catheterization) equal to or below 20%
* patients with cardiac valvular disease
* patients with a spirometry measurement that demonstrates an FEV1/FVC ratio below 60%
* patients with chronic renal failure who require dialysis or
* those who have experienced an allergic reaction to anesthesia in the past
* patients with a history of lung infiltrate on chest X-ray prior to surgery or a history of asthma
* Women who are pregnant are excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

PRIMARY OUTCOMES:
Post-surgical lung function, compliance, tissue oxygenation, and radiographic changes indicative of atelectasis. | During in-patient stay
  Determination if ventilation during surgery improves post-surgical lung function, compliance, tissue oxygenation, and radiographic changes indicative of atelectasis.

CONTACTS AND LOCATIONS:
Overall Officials: Raul Mendoza-Ayala, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora BayCare Medical Center, Green Bay, Wisconsin, United States